CLINICAL TRIAL: NCT04908527
Title: Effect of Walking to the Operating Room on Preoperative Anxiety in Patients Scheduled for Outpatient Laser Therapy for Venous Insufficiency: A Monocentric Randomized Study
Brief Title: Effect of Walking to the Operating Room on Preoperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Claude Hallet, Principal investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-122
Record Dates: First submitted 2021-05-12; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Vein, Varicose
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walk group (Experimental): Patients walked to operating room (OR)
  Interventions: Behavioral: Walking to OR
- Bed group (No Intervention): Patients go to OR while in bed

INTERVENTIONS:
Behavioral: Walking to OR — Patients, after being prepared for the OR, walk to the operating room
  Arms: Walk group

SUMMARY:
The operating room environment can be a source of anxiety for the patient, including in the context of outpatient surgery for which anxiolytic medication is rarely used. This anxiety-induced effect can be reinforced by the patient's lack of active participation.

Some studies have already shown the feasibility of patient walking to the operating room (OR) and advantages this approach(Kojima and Ina 2002; Lack 2016; Nagraj et al. 2006).

Moreover, recovery room complications and pain have also been shown to be greater after varicose vein surgery in patients with significant preoperative anxiety (Scavee et al. 2016).

Therefore, the investigators decided to test the effects of walking to OR for patients admitted for outpatient surgery for varicose vein surgery.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient minimal invasive laser therapy for venous insufficiency

Exclusion Criteria:

* Inpatient surgery
* Invasive surgery
* Need for premedication
* Use of walking aid
* Non-French speaking patient
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Level of anxiety | Preoperatively in the room
  French version of Preoperative Anxiety and Information Scale (APAIS) - Score between 6 (less anxious) and 30 (more anxious)
Level of anxiety | Preoperatively in the room
  Numerical rating scale (NRS) between 0 (= no anxiety) and 10 (=worse anxiety)
Level of anxiety | Preoperatively in front of OR
  Numerical rating scale (NRS) between 0 (= no anxiety) and 10 (=worse anxiety)
Level of anxiety | Before departure of the outpatient unit
  Numerical rating scale (NRS) between 0 (= no anxiety) and 10 (=worse anxiety)

SECONDARY OUTCOMES:
Level of pain | Within 1 hour after admission in the Post Anesthesia Care Unit after surgery
  Numerical rating scale (NRS) between 0 (= no pain) and 10 (=worse pain)
Level of pain | Before departure of outpatient unit
  Numerical rating scale (NRS) between 0 (= no pain) and 10 (=worse pain)
Level of pain | At Day 1
  Numerical rating scale (NRS) between 0 (= no pain) and 10 (=worse pain)
Presence of nausea and vomiting | During the stay in the Post Anesthesia Care Unit after surgery assessed up to 12h
  Yes or No
Presence of nausea and vomiting | During the stay in the outpatient unit after surgery assessed up to 12h
  Yes or no
Presence of nausea and vomiting | at Day 1
  Yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Claude Hallet, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- Centre hospitalier universitaire de Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No